CLINICAL TRIAL: NCT06158672
Title: The Effect of Emotional Freedom Technique on Menopausal Symptoms, Quality of Life and Depression Level: An Experimental Study
Brief Title: The Effect of Emotional Freedom Technique on Menopausal Symptoms, Quality of Life and Depression Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUESRAKARATASOKYAY003
Record Dates: First submitted 2023-11-18; First posted 2023-12-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Menopause
Keywords: Menopause Symptoms; Quality of Life; Depression; Emotional Freedom Technique
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional freedom technique group (Experimental): Emotional freedom technique will be applied to menopausal women in the emotional freedom technique group.
  Interventions: Behavioral: Emotional freedom technique group
- Sham Emotional freedom technique group (Placebo Comparator): Menopausal women in the sham emotional freedom technique group will receive sham emotional freedom technique.
  Interventions: Behavioral: Sham emotional freedom technique group
- Control group (No Intervention): Menopausal women in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Emotional freedom technique group — Menopausal women in the emotional freedom technique group will be administered the emotional freedom technique by the researcher a total of 4 times at one week intervals.
  Arms: Emotional freedom technique group
Behavioral: Sham emotional freedom technique group — Menopausal women in the sham emotional freedom technique group will be administered sham emotional freedom technique by the researcher a total of 4 times with one week intervals.
  Arms: Sham Emotional freedom technique group

SUMMARY:
Emotional freedom technique will be applied to menopausal women. Emotional freedom technique group, sham emotional freedom technique group and control groups each consisted of 35 menopausal women.

DETAILED DESCRIPTION:
Objective: The aim of the study was to determine the effect of emotional freedom technique (EFT) on menopausal symptoms, quality of life and depression level.

Materials and Methods: This randomized controlled trial will be conducted with a total of 105 menopausal women at Fırat Family Health Center and Göztepe Family Health Center between January 2024 and June 2024 (35 EFT, 35 sham, 35 control). EFT and Sham EFT will be applied in the study. Women in the EFT group will receive EFT four times at one week intervals. Women in the Sham EFT group will receive Sham EFT four times with one week intervals. Before the applications, pre-test data will be obtained by filling out the Personal Information Form, Perimenopausal Depression Scale, Menopause Specific Quality of Life Scale and Menopause Symptom Assessment Scale before the application of Emotional Freedom Technique. After the applications, post-test data will be obtained by filling out the Perimenopausal Depression Scale, Menopause Specific Quality of Life Scale and Menopause Symptom Assessment Scale. In addition, the Subjective Units of Experience (SUE) scale will be applied before and after each EFT intervention.

ELIGIBILITY:
Inclusion Criteria:

* A person who has gone through menopause naturally,
* No menstruation for the last one year,
* Literate,
* Not taking Hormone Replacement Therapy,
* No oncologic disease,
* No infection, wound, scar in the tapping areas,
* Women who are able to communicate will be included in the study.

Exclusion Criteria:

* One who has not gone through menopause naturally,
* Illiterate,
* Receiving Hormone Replacement Therapy,
* Women with conditions such as infections, wounds, scars in the tapping areas.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Determining the level of perimenopausal depression | The Perimenopausal Depression Scale will be administered to three groups of menopausal women on day one (first interview).
  The scale was developed to rate the severity of perimenopausal depression symptoms. The scale consists of 12 items and five subscales related to energy, paranoid ideation, irritability, self-esteem, isolation, anxiety, somatic symptoms, sleep disturbance, weight, sexual interest, memory and concentration. All items of the scale are scored between 0 and 4. The lowest score that can be obtained from the scale is 0 and the highest score is 48. An increase in the scale score indicates an increase in depressive symptom status. A score range of 20-24 points indicates mild perimenopausal depression, a score range of 24- 32 points indicates moderate perimenopausal depression requiring treatment, and a score of 32 points and above indicates severe perimenopausal depression requiring treatment.
Determining the level of perimenopausal depression | The Perimenopausal Depression Scale will be administered to three groups of menopausal women at the last interview (after the 4th intervention at one week interval).
  The scale was developed to rate the severity of perimenopausal depression symptoms. The scale consists of 12 items and five subscales related to energy, paranoid ideation, irritability, self-esteem, isolation, anxiety, somatic symptoms, sleep disturbance, weight, sexual interest, memory and concentration. All items of the scale are scored between 0 and 4. The lowest score that can be obtained from the scale is 0 and the highest score is 48. An increase in the scale score indicates an increase in depressive symptom status. A score range of 20-24 points indicates mild perimenopausal depression, a score range of 24- 32 points indicates moderate perimenopausal depression requiring treatment, and a score of 32 points and above indicates severe perimenopausal depression requiring treatment.
Determining quality of life | The Menopause Specific Quality of Life Scale will be administered to three groups of menopausal women on day one (first interview).
  The Menopause Specific Quality of Life Scale assesses the quality of life of menopausal women. The scale consists of 29 Likert-type questions and 4 sub-domains: vasomotor, psychosocial, physical and sexual. The score for each question varies between 1 and 8. In scoring, a score of 1 indicates that the situation was not experienced, a score of 2 indicates that the situation was experienced but not disturbing, and a score between 3-8 indicates the severity of the situation. The score of each sub-domain is obtained by averaging the scores of the items in the sub-domain. A high score on the scale indicates a low quality of life.
Determining quality of life | The Menopause Specific Quality of Life Scale will be administered to three groups of menopausal women at the last interview (after the 4th intervention at one week interval).
  The Menopause Specific Quality of Life Scale assesses the quality of life of menopausal women. The scale consists of 29 Likert-type questions and 4 sub-domains: vasomotor, psychosocial, physical and sexual. The score for each question varies between 1 and 8. In scoring, a score of 1 indicates that the situation was not experienced, a score of 2 indicates that the situation was experienced but not disturbing, and a score between 3-8 indicates the severity of the situation. The score of each sub-domain is obtained by averaging the scores of the items in the sub-domain. A high score on the scale indicates a low quality of life.
Assessment of menopausal symptoms | The Menopausal Symptoms Rating Scale will be administered to three groups of menopausal women on day one (first interview).
  The Menopausal Symptoms Rating Scale measures the severity of menopausal symptoms. In the Likert-type scale consisting of a total of 11 items including menopausal complaints, there are "0= None", "1= Mild", "2= Moderate", "3= Severe" and "4= Very severe" options for each item. The total score of the scale is calculated based on the scores given for each item. The lowest score that can be obtained from the scale is 0 and the highest score is 44. An increase in the total score indicates an increase in the severity of the complaints experienced. The scale consists of three subscales (Somatic Complaints Subscale, Psychological Complaints Subscale, Urogenital Complaints Subscale).
Assessment of menopausal symptoms | The Menopause Symptoms Assessment Scale will be administered to three groups of menopausal women at the last interview (after the 4th intervention at one week interval).
  The Menopausal Symptoms Rating Scale measures the severity of menopausal symptoms. In the Likert-type scale consisting of a total of 11 items including menopausal complaints, there are "0= None", "1= Mild", "2= Moderate", "3= Severe" and "4= Very severe" options for each item. The total score of the scale is calculated based on the scores given for each item. The lowest score that can be obtained from the scale is 0 and the highest score is 44. An increase in the total score indicates an increase in the severity of the complaints experienced. The scale consists of three subscales (Somatic Complaints Subscale, Psychological Complaints Subscale, Urogenital Complaints Subscale).
Determining the level of anxiety | The Subjective Units of Experience (SUE) scale will be administered to three groups of menopausal women on day one (first interview).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the first interview, all menopausal women in all three groups will be administered the SUE (second measure).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | Seven days after the first interview, all menopausal women in all three groups will be administered the SUE (third measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the third measurement, all menopausal women in all three groups will be administered the SUE (fourth measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | Seven days after the fourth measurement, all menopausal women in all three groups will be administered the SUE (fifth measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the fifth measurement, all menopausal women in all three groups will be administered the SUE (sixth measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | Seven days after the sixth measurement, all menopausal women in all three groups will undergo the SUE (seventh measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.
Determining the level of anxiety | One hour after the seventh measurement, all menopausal women in all three groups will be administered the SUE (eighth measurement).
  Subjective Units of Experience (SUE) will be applied to determine the anxiety level of menopausal women. The SUE is used to determine the intensity of one's emotions at the beginning and end of the therapy. The scale is scored between -10 and +10, with negative numbers indicating negative/unpleasant experiences and positive numbers indicating positive/pleasant experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Esra KARATAŞ OKYAY, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; Zeliha ÖZŞAHİN, PhD, Study Director — Inonu University; Çiğdem KARAKAYALI AY, PhD, Study Director — Kahramanmaras Sutcu Imam University; Sinem GÜVEN SANTUR, Master, Study Director — Inonu University
Locations (2):
- Turkey (Türkiye) (2):
  - Firat Family Health Center, Malatya
  - Göztepe Family Health Center, Malatya

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Background] Mehdipour A, Abedi P, Ansari S, Dastoorpoor M. The effectiveness of emotional freedom techniques (EFT) on depression of postmenopausal women: a randomized controlled trial. J Complement Integr Med. 2021 May 19;19(3):737-742. doi: 10.1515/jcim-2020-0245. eCollection 2022 Sep 1. PMID 34013673
- See also: Description citation link — https://pubmed.ncbi.nlm.nih.gov/34013673/